CLINICAL TRIAL: NCT04321148
Title: Prospective Randomized Study Comparing Impella Support Plus Optimal Medical Care Versus Optimal Medical Care Alone in Patients at High Risk for Contrast-induced Nephropathy Undergoing Elective Percutaneous Revascularization
Brief Title: Protect Kidney Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: Profil Clinical Trials Coordination GmbH (Unknown); Abiomed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-018
Record Dates: First submitted 2020-03-16; First posted 2020-03-25 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Induced Acute Kidney Injury; High-risk Percutaneous Coronary Intervention
Keywords: induced acute kidney injury; high-risk percutaneous coronary intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard of care PCI (Other)
  Interventions: Procedure: standard of care PCI
- Impella-protected PCI (Experimental)
  Interventions: Procedure: Impella-protected PCI

INTERVENTIONS:
Procedure: standard of care PCI — optimal medical care PCI
  Arms: standard of care PCI
Procedure: Impella-protected PCI — Impella-protected PCI
  Arms: Impella-protected PCI

SUMMARY:
This trial is a randomized, controlled, open-label, parallel study. Patients at high risk for contrast induced acute kidney injury (CI AKI) and planned high-risk percutaneous coronary intervention (PCI) will be randomized to receive optimal medical care for the prevention of CI AKI with periprocedural hydration either in combination with or without use of an Impella device during PCI. Renal function will be assessed over 6 months, potential complications (in particular bleeding and access site complications) over one month. Effects of device-assisted PCI on pathways for salt and water handling, as well as on kidney oxygenation will be detected by sequential sampling of blood and urine as well as detection of magnetic resonance imaging indicative of blood kidney oxygenation (BOLD MRI).

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent obtained before any trial-related activities.
2. Patients aged 18-85 years (both inclusive) with clinical indication for coronary angiogram with potential high-risk PCI
3. Patients at high risk for contrast induced acute kidney injury as indicated by a preliminary Mehran Score ≥ 10 (contrast media volume is assumed to be < 100 ml)

Exclusion Criteria:

1. Previous participation in this trial. Participation is defined as randomized.
2. Patients with contraindications to use of an Impella heart pump (mural thrombus in the left ventricle; presence of a mechanical aortic valve or aortic valve stenosis (equivalent orifice area of 1.5 cm2 or less); moderate to severe aortic insufficiency (echocardiographic assessment graded as ≥ +2); in whom severe peripheral arterial disease precluding placement of an Impella system)
3. Patients where hemodynamic support is deemed potentially required for PCI as assessed by at least one physician
4. Patients needing emergency percutaneous coronary intervention (e.g. STEMI patients)
5. Patients with acute cardiogenic shock indicated by one of the following:

   1. Systolic blood pressure < 90mmHg over 30 minutes or inotropic support needed to maintain blood pressure targets.
   2. Killip class III & IV
   3. MCS already in place to maintain blood pressure and organ perfusion
6. Patients with on-going resuscitation
7. Unwitnessed cardiac arrest OR ≥30 minutes of CPR prior to screening OR any impairment in mental status, cognition, or any global or focal neurological deficit
8. Patients on mechanical ventilation.
9. Patients diagnosed with AKI within the last seven days prior to screening or incipient AKI. (In cases, where AKI cannot be ruled out as a cause for elevated serum creatine, a rise or fall above 30% of a second serum creatinine measurement obtained within 12 to 24 hours is indicative of AKI)
10. Patients with an eGFR < 20 ml/min/1.73 m²
11. Suspected or known pregnancy
12. Patients with comorbidity that in the Investigator's opinion would limit life expectancy to less than 6 months
13. Patients with other medical, social, or psychological problems that, in the opinion of the Investigator, preclude them from undergoing Impella-protected PCI or the study-related procedures, evaluations, and follow-up.
14. Patients with severe anemia as indicated by hemoglobin concentrations < 8.5 g/dl at the time of screening.
15. Patients who were exposed to contrast media in the last seven days prior to the time of screening
16. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
17. Participation in the active treatment or follow-up phase of another clinical study of an investigational drug or device which has not reached its primary end point.

Patients with contraindications against MRI-procedures (e.g. patients with pacemakers) are eligible for the study but will not participate in the BOLD-MRI assessment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2020-01-24 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of Contrast-induced acute kidney injury (CI-AKI) | 2 days after PCI
  Incidence rate of AKI (Acute Kidney Injury Criteria 1-3) over 2 days after PCI

SECONDARY OUTCOMES:
Change in eGFR | at day 1 and day 3 from baseline (pre-PCI)
Incidence of acute kidney injury (AKIN Criteria 1-3) | over 3 days after PCI
Incidence of dialysis | up to 6 months after PCI
  Incidence of dialysis during hospitalization and over 6 months after PCI
Incidence of re-hospitalization for renal dysfunction | 30 days and up to 6 months after PCI
  Incidence of re-hospitalization for renal dysfunction over 30 days and 6 months after PCI
Mortality | up to 6 months after PCI
  Mortality during hospital stay and over 6 months after PCI
Length of hospital stay | up to 3 days after PCI

CONTACTS AND LOCATIONS:
Locations (1):
- Heinrich-Heine-University, Div. of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided